CLINICAL TRIAL: NCT03528122
Title: The Safety and Efficacy of Using Amniotic Membrane for Closure of Recurrent Macular Hole
Brief Title: Amniotic Membrane for Recurrent Macular Hole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hossam Mohamed Moharram, Assistant Professor of Ophthalmology, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63 2/2018
Record Dates: First submitted 2018-04-21; First posted 2018-05-17 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Macula Hole; Retinal Detachment; Myopic Macular Degeneration
Keywords: amniotic membrane; retinal detachment; Myopic; macular hole; internal limiting membrane
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment; Myopia

STUDY DESIGN:
Intervention Model Description: Individuals with recurrent macular hole associated retinal detachment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent opened macular hole (Experimental): Pars plana vitrectomy with internal limiting membrane peel if not peeled in the first surgery and application of amniotic membrane graft
  Interventions: Procedure: Recurrent opened macular hole

INTERVENTIONS:
Procedure: Recurrent opened macular hole — pars plana vitrectomy + internal limiting membrane peeling + Amniotic membrane graft placement over the hole + intraocular tamponade

SUMMARY:
Macular hole surgery were tried by different surgeons using many techniques with different successes but still there were many recurrences. In this study the investigators try to close these distinct types including recurrent holes using pre-prepared amniotic membrane.

DETAILED DESCRIPTION:
It is an interventional study of using amniotic membrane graft for closure of macular hole associated retinal detachment in patient who had a previous failed macular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with history of opened macular hole after previous pars plana vitrectomy and internal limiting membrane (ILM) peeling for treatment of myopic macular hole were included.
* Opened holes after 1 month of the surgery.
* Myopic macular holes only were included (Refraction of more than _6 D and/or axial length of more than 26 mm).

Exclusion Criteria:

* All other causes of macular hole (traumatic and idiopathic)
* Patients with diseases that can affect visual outcome (Diabetic retinopathy, choroidal neovascularization, age-related macular disease and advanced glaucoma patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical restoration of macular hole closure | 6 months
  Closure of the macular hole

SECONDARY OUTCOMES:
Functional restoration after closure of the macular hole | 6 months
  Improvement of the best corrected visual acuity (BCVA)
Functional restoration after closure of the macular hole | 6 months
  Any improvement of the waves in the electrophysiological (ERG) study.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia UNiversity hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided